CLINICAL TRIAL: NCT00032305
Title: A Phase I, Dose-Escalation, Pilot Study of Visilizumab in Patients With Severe Ulcerative Colitis That is Refractory to Corticosteroids
Brief Title: Research Study in Patients With Severe Ulcerative Colitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Facet Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 291-406
Record Dates: First submitted 2002-03-14; First posted 2002-03-18 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Ulcerative Colitis
Keywords: Colitis; Gastrointestinal Disease; Digestive System Disease; Intestinal Disease; Colonic Disease
MeSH Terms: conditions — Colitis, Ulcerative; Colitis; Gastrointestinal Diseases; Digestive System Diseases; Intestinal Diseases; Colonic Diseases | interventions — visilizumab

INTERVENTIONS:
Drug: Visilizumab

SUMMARY:
The purpose of the study is to evaluate an intravenous (by injection) investigational medication to treat severe ulcerative colitis refractory to steroid therapy. The research is being conducted at up to 8 clinical research sites in the US and is open to both men and women ages 18 to 70 years old. Participants in the study will have a number of visits to a research site. All study-related care and medication is provided to qualified participants at no cost: this includes all visits, examinations and laboratory work.

DETAILED DESCRIPTION:
A Phase I, dose-escalation, pilot study designed to obtain safety and tolerability data on visilizumab administered to patients with severe ulcerative colitis that has failed to respond to steroid therapy. Patients who are currently receiving IV corticosteroids, but whose disease has not responded after at least 5 days of this therapy, will be eligible for the study.

ELIGIBILITY:
1. A diagnosis of ulcerative colitis verified by colonoscopy or barium enema performed within 36 months prior to study entry.
2. Active disease despite ongoing treatment with steroids

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2002-03; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California, San Francisco, California
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - The University of Chicago Medical Center, Chicago, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - Mount Sinai School of Medicine, New York, New York
  - University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Plevy S, Salzberg B, Van Assche G, Regueiro M, Hommes D, Sandborn W, Hanauer S, Targan S, Mayer L, Mahadevan U, Frankel M, Lowder J. A phase I study of visilizumab, a humanized anti-CD3 monoclonal antibody, in severe steroid-refractory ulcerative colitis. Gastroenterology. 2007 Nov;133(5):1414-22. doi: 10.1053/j.gastro.2007.08.035. Epub 2007 Aug 21. PMID 17920064